CLINICAL TRIAL: NCT03174730
Title: Investigating a Technology Delivered Growth Mindset Intervention for Smoking Cessation.
Brief Title: Mindset Intervention for Nicotine Dependence
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8545
Record Dates: First submitted 2017-04-19; First posted 2017-06-02 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Psychology, Social; Smoking Cessation; Smoking (Tobacco) Addiction
Keywords: smoking; smartphone; technology; addiction
MeSH Terms: conditions — Smoking Cessation; Smoking; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: All participants will gain access to SmartQuit, a smartphone based app with tools for quitting smoking. In order to test whether the growth mindset intervention is effective, smokers will be randomly assigned to either an experimental group, where they will additionally get growth mindset content or to a control group.
Who Masked: Participant
Masking Description: In order to control for expectancy or placebo effects, participants will be told that the study is designed to test the method of delivery of content (email vs. smartphone). They will not be aware that one group is getting something extra that the control group is not getting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth mindset (Experimental): In addition to SmartQuit (the app), study participants will receive the content in the form on one growth mindset tip (sent in an email) per day starting on the first day of the study. Email exercises will be sent out every 3 days and there are a total of 8 emails.
  Interventions: Behavioral: Growth Mindset; Behavioral: SmartQuit
- Control (Other): Participants will get SmartQuit, but not the growth mindset intervention.
  Interventions: Behavioral: SmartQuit

INTERVENTIONS:
Behavioral: Growth Mindset — The intervention is aimed at creating more flexible thinking about addiction to tobacco. Participants will be sent tips by email to help foster the belief that people can overcome addiction to smoking.
  Arms: Growth mindset
Behavioral: SmartQuit — This is an Acceptance and Commitment Therapy based intervention designed a smoking cessation smartphone application.

SUMMARY:
This study evaluates a new digitally delivered mindset based intervention in addition to a smartphone application (app) for smoking cessation. Participants will be provided an app (SmartQuit) that teaches them skills to quit, and will be randomly assigned to either receive a growth mindset intervention or to a control group.

DETAILED DESCRIPTION:
Want to quit smoking? Welcome to the MIND Study, conducted by researchers at Seattle's Fred Hutchinson Cancer Research Center.

Join now to get a smartphone app-based quit smoking program that includes:

* Personalized plans for quitting
* Help with dealing with urges to smoke
* Information on nicotine withdrawal
* Help staying motivated
* Tracking progress with quitting
* A certificate of completion once you complete the program
* Scientifically-based information on quit medications

The MIND study gives you all these and more to help you quit smoking and live a happier, healthier life. For more information, visit mind.fredhutch.org.

ELIGIBILITY:
Inclusion Criteria:

(1) age 18 or older, (2) smokes at least five cigarettes daily for at least past 12 months, (3) wants to quit in the next 30 days, (4) interested in learning skills to quit smoking, (5) resides in US, (6) has at least daily access to their own smartphone, (7) knows how to login and download a smartphone application from their smartphone, (8) willing and able to read in English, (9) not participating in other smoking cessation interventions (including our other intervention studies). To increase follow-up retention, eligibility criteria also include: (10) willing to complete one follow-up survey, (11) provide email, phone, and mailing address.

Exclusion Criteria:

Opposite of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Engagement with smoking cessation program | 2 months
  Number of times the smoking cessation app is opened, number of days logged in to smoking cessation app
Cessation of smoking | 2 months
  30 day point prevalence abstinence [i.e. no smoking for the past 30 days]

SECONDARY OUTCOMES:
Cessation of smoking | 2 months
  7 day point prevalence abstinence [i.e. no smoking in past 7 days]

OTHER OUTCOMES:
Mediation of engagement | 2 months
  The effect of mindset intervention on engagement outcomes will be mediated by change in mindset.
Mediation of cessation | 2 months
  The effect of mindset intervention on cessation outcomes will be mediated by change in mindset.
Moderation by mindset | 2 months
  Mindset at baseline moderates the treatment effect such that engagement and cessation outcomes improve more for those smokers who start the study with a fixed mindset.
Number of cigarettes smoked per day (reduction) | 2 months
  Test to see whether there is reduced smoking in one arm compared to the other.

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sridharan V, Shoda Y, Heffner J, Bricker J. A Pilot Randomized Controlled Trial of a Web-Based Growth Mindset Intervention to Enhance the Effectiveness of a Smartphone App for Smoking Cessation. JMIR Mhealth Uhealth. 2019 Jul 9;7(7):e14602. doi: 10.2196/14602. PMID 31290404